CLINICAL TRIAL: NCT02260167
Title: Effective Treatment of Alzheimer's and Dementia With the MIND Protocol
Brief Title: Treatment of Alzheimer's and Dementia With the Metabolism, Infections, Nutrition, Drug Elimination (MIND) Protocol
Acronym: MIND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Practitioners Alliance Network (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PAN-ALZ002
Record Dates: First submitted 2014-10-05; First posted 2014-10-09 (Estimated); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Alzheimer's Disease; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment with MIND (Experimental)
  Interventions: Other: A mix of natural treatments and medications

INTERVENTIONS:
Other: A mix of natural treatments and medications
  Other Names: MIND Protocol

SUMMARY:
Treating with measures that may improve metabolic functioning of neurons in an integrated protocol

DETAILED DESCRIPTION:
Most organ failure results in modest drops in function until over 50% of function is lost. At a certain point, even modest drops in physiologic activity result in dramatic drops in clinical function. Though less homogeneous than in other organs, clinical experience and the literature suggests a similar process occurs in the brain. The hypothesis is that by using an integrated protocol to, essentially, "tune up" neuronal function, a 5-10 % improvement in metabolic functioning may translate to significant improvement in clinical functioning. This tune-up will include "MIND":

M- Metabolism-- optimizing hormonal function I- Infections-- looking for and eliminating N- Nutritional and herbal support D- Drugs- Weaning subjects off unneeded medications

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of Alzheimer's and/or dementia with an MMSE score over 12 or being ambulatory and able to travel outside the home with assistance.
* Must have a caregiver living with them.

Exclusion Criteria:

* Overt progressive and severe causes of secondary dementia such as metastatic brain cancers, or severe overt infectious encephalopathies or severe autoimmune illness.
* Also, severe life threatening illnesses which would make them unlikely to be alive after 6-12 months

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2014-09 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 6 months
  Looking to see what percent of patients show improvement

SECONDARY OUTCOMES:
Mini Mental Status Exam (MMSE) | 6 months
Alzheimer's Disease Assessment Scale- Activities of Daily Living (ADAS-ADL) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- PAN, Kailua, Hawaii, United States

IPD SHARING:
Plan to Share IPD: No